CLINICAL TRIAL: NCT03283839
Title: Consequences of Temporomandibular Disorder on Balance Control
Acronym: DAM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-A01317-44
Record Dates: First submitted 2017-05-19; First posted 2017-09-14 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Temporomandibular Disorder; Pathophysiology; Therapy
Keywords: Temporo-mandibular dysfunction; Balance control; Orientation function
MeSH Terms: conditions — Temporomandibular Joint Disorders; Orientation, Spatial

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Temporomandibular disorder (Other)
  Interventions: Diagnostic Test: Posturography
- Without temporomandibular disorder (Other)
  Interventions: Diagnostic Test: Posturography

INTERVENTIONS:
Diagnostic Test: Posturography — Evaluation of postural control and of orientation function
  Other Names: Orientation perception

SUMMARY:
To evaluate the effects of the temporomandibular disorder (TMD) and its therapeutic care on postural control in somato-sensory and visual sensitization compared to control subjects matched on age, sex and lifestyle.

Parameters will be estimated by measures realized before the therapeutic care of the TMD (T0), then 2, 3 and 5 months after the starting care, both in TMD patients and control subjects. To evaluate also the effects of the TMD and its therapeutic care on balance control in various contexts of multi-sensory stimulation, orientation function, pain and tinnitus.

DETAILED DESCRIPTION:
Primary objective: to evaluate the effects of the temporomandibular disorder (TMD) and its therapeutic care on postural control in somato-sensory and visual sensitization compared to control subjects matched on age, sex and lifestyle.

ELIGIBILITY:
Inclusion Criteria:

* Patient group: TMD patients, care: occlusal splint therapy, behavioral advices
* Control group: matched with TMD patients (age, sex, lifestyle).

Exclusion Criteria:

* Patient group: treatment generating secondary effects in postural control (psychotrop, antidepressor, antihypertensive drugs); osteoarticular pathologies and recent trauma (< 4 months); vertigo and dysequilibrium (< 6 months), whiplash
* Control group: id. and TMD.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-06-19 (Actual); Primary Completion 2019-02-25 (Estimated); Study Completion 2020-06-25 (Estimated)

PRIMARY OUTCOMES:
Postural control (before care for patients) | At inclusion (before care for patients) (first evaluation)
  Postural control is evaluate by the average of condition 5 and 6 of the sensory organisation test (SOT) measured on Equitest plateform.
Postural control (during care for patients) | 2 months after the first evaluation
  Postural control is evaluate by the average of condition 5 and 6 of the sensory organisation test (SOT) measured on Equitest plateform.
Postural control (during care for patients) | 3 months after the first evaluation
  Postural control is evaluate by the average of condition 5 and 6 of the sensory organisation test (SOT) measured on Equitest plateform.
Postural control (during care for patients) | 5 months after the first evaluation
  Postural control is evaluate by the average of condition 5 and 6 of the sensory organisation test (SOT) measured on Equitest plateform.

SECONDARY OUTCOMES:
Balance function | T0 and 2,3 and 5 months after the first evaluation
  Length and surface covered by the foot pressure center are measured
Orientation function | T0 and 2,3 and 5 months after the first evaluation
  Orientation is evaluated by the angle between the direction (of the gravity or of a part of his body) indicated by the subject and the real direction. It is evaluated with the road and frame test.
Pain | T0 and 2,3 and 5 months after the first evaluation
  Visual Analog Scale (1 to 10)
Tinnitus | T0 and 2,3 and 5 months after the first evaluation
  Questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de NANCY, Nancy, France

IPD SHARING:
Plan to Share IPD: No